CLINICAL TRIAL: NCT05368376
Title: Is Labetalol More Effective Than Metoprolol for Controlled Hypotensive Anesthesia During Endoscopic Nasal Surgeries? A Randomized Clinical Trial.
Brief Title: Is Labetalol More Effective Than Metoprolol for Controlled Hypotensive Anesthesia During Endoscopic Nasal Surgeries?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DTH: 22001
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hypotension Drug-Induced
Keywords: controlled hypotension; endoscopic nasal surgery; labetalol; metoprolol
MeSH Terms: conditions — Hypotension | interventions — Labetalol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (n=30) (Active Comparator): Labetalol group
  Interventions: Drug: Labetalol Hydrochloride Oral Tablet
- Group M (n=30) (Active Comparator): Metoprolol group
  Interventions: Drug: Metoprolol Tartrate Oral Tablet

INTERVENTIONS:
Drug: Labetalol Hydrochloride Oral Tablet — Labetalol 200 mg
  Other Names: Labipress tablets
  Arms: Group L (n=30)
Drug: Metoprolol Tartrate Oral Tablet — Metoprolol 100 mg
  Other Names: Betaloc tablets
  Arms: Group M (n=30)

SUMMARY:
Background: Mucosal bleeding is the most frequent complication with endoscopic nasal surgeries, as it interferes with the optimal visualization of the intranasal anatomy, leading to increased complications, operation duration, and blood loss. There are several pharmacological techniques for the appropriate control of intraoperative bleeding.

Objectives: To compare the safety and efficacy of oral labetalol versus oral metoprolol as a premedication for controlled hypotensive anesthesia during endoscopic nasal surgeries.

Patients and Methods: This is a randomized, double-blind, phase four, comparative clinical trial; carried out on 60 patients, who were candidates for endoscopic nasal surgeries under general anesthesia at our hospital. Patients were randomly allocated into two equal groups; group L, received oral labetalol, and group M, received oral metoprolol.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 50 years
* Body Mass Index (BMI) ≤ 35 kg/m2

Exclusion Criteria:

* ASA physical status > II
* Age < 21 years or > 50 years
* Pregnant women
* Breastfeeding
* Bronchial asthma
* Chronic obstructive pulmonary disease
* Hypertension
* Ischemic heart disease
* Rheumatic heart disease
* Heart failure
* Heart block
* Sick sinus syndrome
* Sinus bradycardia
* Chronic hypotension
* Anemia (Hb < 10 g/dl)
* Renal or hepatic dysfunction
* Central nervous system disease
* Bleeding diathesis
* Diabetes Mellitus
* Allergic fungal sinusitis
* Patients on beta-blockers, tricyclic antidepressants, alcohol or drug abuse, anticoagulation therapy, agents influencing the autonomic nervous system
* Patients using pacemakers
* Allergy to the study drugs
* Any contraindication of oral intake

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Mean and Standard deviation of Blood loss (ml)(mean±SD) | 30 minutes after the end of surgery
  Amount of blood loss at the end of surgery

SECONDARY OUTCOMES:
Mean and Standard deviation of Sevoflurane concentration (%)(mean±SD) | 30 minutes after the end of surgery
  Concentration of sevoflurane used during surgery
Mean and Standard deviation of Heart rate (beat/min.)(mean±SD) | 30 minutes after the end of surgery
  Before premedication (T_B), 2 hours after premedication (T0), 1 minute after induction of anesthesia (T1), at 15 (T15), 30 (T30), 45 (T45), 60 (T60), 75 (T75) minutes after induction of anesthesia, at post anesthesia care unit (T_PACU)
Mean and Standard deviation of Mean Blood Pressure (mmHg)(mean±SD) | 30 minutes after the end of surgery
  Before premedication (T_B), 2 hours after premedication (T0), 1 minute after induction of anesthesia (T1), at 15 (T15), 30 (T30), 45 (T45), 60 (T60), 75 (T75) minutes after induction of anesthesia, at post anesthesia care unit (T_PACU)
Number of participants and Percentage of Drug-related side effects | 30 minutes after the end of surgery
  Number of participants and Rate of: Bradycardia, Hypotension, Dysrhythmia, Bronchospasm, and Postoperative nausea and vomiting (PONV)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt